CLINICAL TRIAL: NCT03139474
Title: Impact of Gonadotrophin Releasing Hormone Analogues on Oocyte and Embryo Quality in Intracytoplasmic Sperm Injection Cycles.
Brief Title: Impact of Gonadotrophin Releasing Hormone Analogues on Oocyte and Embryo Quality
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Traiza Helal, Dr., Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYY
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- agonist group (Active Comparator): Triptorelin at a dose 1 milligram per day from the midluteal phase of the cycle preceding the treatment cycle to day 2 of the cycle then 0.5 milligram of triptorelin will be used during the period of stimulation.
  Interventions: Drug: Gonadotropin-Releasing Hormone Analogue
- antagonist group (Active Comparator): •Multiple dose Gonadotrophin releasing hormone antagonist regimen will be used for ovarian stimulation 0.25 microgram per day cetrorelix will be administered from the 6th day of ovarian stimulation or from the presence of follicle 14 millimeter diameter .
  Interventions: Drug: Gonadotropin releasing hormone antagonist

INTERVENTIONS:
Drug: Gonadotropin-Releasing Hormone Analogue — Triptorelin at a dose 1 mg per day from the midluteal phase of the cycle preceding the treatment cycle to day 2 of the cycle then 0.5 milligram of triptorelin will be used during the period of stimulation.
  Arms: agonist group
Drug: Gonadotropin releasing hormone antagonist — antagonist group :Multiple dose gonadotrophin-releasing hormone antagonist regimen will be used for ovarian stimulation 0.25 microgram per day cetrorelix will be administered from the 6th day of ovarian stimulation or from the presence of follicle 14 millimeter diameter .We will give them gonadotrophin for 5 days , Triggering by Human Chorionic Gonadotrophin will be administered for each group when size of follicle reach > 17 millimeter .Oocytes will retrieved by transvaginal ultrasound , 34-36 hours after Human Chorionic Gonadotrophin administration .
  Arms: antagonist group

SUMMARY:
The first In-Vitro Fertilization cycles were performed in natural unstimulated cycles. Today gonadotrophins are administered to induce multiple follicular development and controlled ovarian hyperstimulation. During ovarian stimulation gonadotrophin-releasing hormone analogues are co-administered in order to prevent premature luteinizing hormone surges. Premature luteinizing hormone surges are observed in about 20% of stimulated cycles without using gonadotrophin-releasing hormone analogues .

Avoiding the adverse effects of elevated luteinizing hormone levels, first gonadotrophin-releasing hormone agonist analogues were used to supplement the gonadotrophin stimulation. The continuous administration of gonadotrophin-releasing hormone agonists causes gonadotrophin suppression through down-regulation and desensitization of the gonadotrophin-releasing hormone receptors in the pituitary gland after an initial short period of gonadotrophin hypersecretion .

Gonadotrophin-releasing hormone antagonists (cetrorelix and ganirelix) cause immediate and rapid gonadotrophin suppression by competitive antagonism of the gonadotrophin-releasing hormone receptor in the pituitary without an initial period of gonadotrophin hypersecretion. Several advantageous effects of cetrorelix were established , and these effects seemed to be independent from the type of antagonist used for luteinizing hormone-suppression.The quality of oocytes and developing preembryos is one of the most relevant factors determining the success of an In-Vitro Fertilization treatment. As ovarian stimulation protocol is one of the eligible factors during an In-Vitro Fertilization treatment, its embryo quality influencing effects are necessary to know.

ELIGIBILITY:
Inclusion Criteria:

1. Unexplained infertility.
2. Tubal factor. Included treated hydrosalpinx and pyosalpinx
3. first cycle .
4. Body mass index: 18-29.
5. Follicle stimulating hormone not more than 14 , E2 not more than 80 and Antimullerian hormone >1.
6. Antral follicular count: more than 5 follicles in one ovary.
7. combined factors .
8. Normal male semen analysis: Mild male factor: concentrations 10 million - 20 million sperm/ml. Moderate male factor : concentrations 5 million - 10 million sperm/ml.

Exclusion Criteria:

1. Patients with Endometriosis.
2. Azoospermic male.
3. Body mass index more than 29.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
number of maturated oocyte and good quality embryoes | 14 days

SECONDARY OUTCOMES:
clinical pregnancy outcome | 6 weeks

IPD SHARING:
Plan to Share IPD: Undecided